CLINICAL TRIAL: NCT06355505
Title: Process of Emergence and Implementation of Advanced Practice Nursing in France
Acronym: PEIPA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PREPS-21-0098
Record Dates: First submitted 2024-03-25; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Nurse's Role
Keywords: advanced practice nursing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Graduate APNs: 700 participants who hold the state diploma of advanced practice nurse and have been practising for more than 6 months as an APN in a hospital structure, in a health establishment in primary care or via a liberal activity in primary care
- 3 consecutive classes of advanced practice students: 900 participants recruited during the 2nd year of training from 3 consecutive classes of students

SUMMARY:
Longitudinal, observational research with a mixed quantitative (by questionnaires) and qualitative (by interviews and observations) approach, multidisciplinary, among Advanced Practice Nurses (APNs) already graduated and 3 consecutive classes of advanced practice students who will be followed annually during their implementation as APN until the last year of the study. The questionnaires will focus on APN scope of practice evolution, economical analysis and geographical distribution of APN. The ethnographical approach will assess APN settlements and relation with healthcare colleagues and patients.

DETAILED DESCRIPTION:
For 40 years, France has faced an increase in demand for care. At the same time, it faces problems of scarcity and unequal geographical distribution of human resources in health. Recent projections by the Ministry of Health predict a decline in French medical density over the next few years, which would more particularly concern the provision of care in private general practice. According to the Organisation for Economic Co-operation and Development (OECD), this development raises fears that the already significant spatial inequalities in staffing will be exacerbated. Another key player are nurses (state registered nurses), who remain insufficiently numerous and unevenly distributed, although their density is increasing in France as in most OECD countries. The WHO (World Health Organization) recommends strengthening the attractiveness of their profession and rethinking professional boundaries in order to foster cooperation with the medical professions.

In France, the framework of practice of some state registered nurses has evolved within the framework of programs aimed at developing the delegation of tasks (cooperation protocols, e.g. Asalé device) and coordinated practice (health homes, health centers). In addition, in 2018, the regulatory framework for advanced practice nursing was created with a dual objective: to improve access to care and the quality of patient pathways. A specific 2-year master's degree course is currently provided by 24 universities. To date, there are 2400 APNs and 700 graduate each year.

Amendment 9 relating to the APN exercise (2023) sets the financial valuation of the advanced practice nursing activity (PAI packages). A pilot study conducted by Julie Devictor et al from 2019 to 2021 showed that among the APNs of the two 1st cohorts, 20% work in primary care (mixed activity APN/state registered nurses majority), 50% in health facilities and 30% do not practice as APNs. Obstacles and levers to the implementation of advanced practice are identified in the international literature. The study hypothesize that there are also some in France, which it is necessary to identify in the context of the health system.

ELIGIBILITY:
Inclusion criteria :

For the questionnaires :

* be enrolled in the 2nd year (semester 3 or 4) in one of the 24 universities offering the State Diploma of Advanced Practice Nursing, regardless of the mention between 2024 and 2026
* be the holder of the state APN diploma at the beginning of the study (year 2024)

For case studies:

- hold the state diploma of Advanced Practice Nurse and have been practicing for more than 6 months as an APN in a hospital structure, in a health facility in primary care or via a liberal activity in primary care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 700 participants recruited among graduate APNs 900 participants recruited during the 2nd year of training from 3 consecutive student classes i.e. 1600 participants in total
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Factors influencing the effective implementation of advanced practice nursing in France in primary care and health facilities | 48 months
  The explanatory variables to be studied will be selected from data from the literature related to the implementation of advanced practice and the obstacles and levers identified internationally.

SECONDARY OUTCOMES:
Mapping of APNs in France with socio-demographic data | 48 months
  Socio-demographic data includes : seniority, professional background, training path, motivations and expectations, access to training, financing studies, diplomas, mode and place of practice, position held, mention, quantification of activity in advanced practice (patients, number of physicians who have signed the organizational protocols, remuneration) and scope of practice / missions carried out (clinical, education, research, leadership, professional development, consultation).
Definition by the APN of its role and missions | 48 months
Implementation and dissemination of the APN practice in the territory according to the context of practice (community care, hospital) | 48 months
  Assessement of the APN scope of practice with an approach internationally validated and used
Identification of potential impact dimensions of Advanced Practice Nursing | 48 months
  Formulation of hypotheses on the extent of these impacts in the following main directions: quality of care and services provided for patients (screening, prevention, follow-up), efficiency of care pathways (medical, specialized and hospital recourse), productivity according to modes and structures of practice.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Devictor, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Beaujon hospital, Clichy, France

IPD SHARING:
Plan to Share IPD: No